CLINICAL TRIAL: NCT03276962
Title: Efficacy, Safety and Immunogenicity Study of GSK Biologicals' Candidate Malaria Vaccine (SB257049) Evaluating Schedules With or With-out Fractional Doses, Early Dose 4 and Yearly Doses, in Children 5-17 Months of Age
Brief Title: Efficacy, Safety and Immunogenicity Study of GSK Biologicals' Candidate Malaria Vaccine (SB257049) Evaluating Schedules With or Without Fractional Doses, Early Dose 4 and Yearly Doses, in Children 5-17 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204889; 2016-000290-20 (EudraCT Number)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Malaria
Keywords: falciparum, efficacy; RTS,S/AS01; malaria vaccine; safety; Malaria; immunogenicity; infants
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine; Rabies Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- R012-20 Group (Experimental): Participants will receive a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2 and at Month 20.
  Interventions: Biological: RTS,S/AS01E (Full dose)
- R012-14-mD Group (Experimental): Participants will receive a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2 and yearly full doses at Month 14, Month 26 and Month 38.
  Interventions: Biological: RTS,S/AS01E (Full dose)
- Fx012-14-mFxD Group (Experimental): Participants will receive a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 2 and yearly fractional doses at Month 14, Month 26 and Month 38.
  Interventions: Biological: RTS,S/AS01E (Full dose); Biological: RTS,S/AS01E (1/5th dose)
- Fx017-mFxD Group (Experimental): Participants will receive a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 7 and yearly fractional doses at Month 20 and Month 32.
  Interventions: Biological: RTS,S/AS01E (Full dose); Biological: RTS,S/AS01E (1/5th dose)
- Control Group (Experimental): Participants will receive rabies vaccine at Month 0, Month 1 and Month 2.
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: RTS,S/AS01E (Full dose) — Participants will receive intramuscular injection of RTS,S/AS01E (full dose: 0.5 ml).
  Arms: Fx012-14-mFxD Group; Fx017-mFxD Group; R012-14-mD Group; R012-20 Group
Biological: RTS,S/AS01E (1/5th dose) — Participants will receive intramuscular injection of RTS,S/AS01E (1/5th dose: 0.1 ml).
  Arms: Fx012-14-mFxD Group; Fx017-mFxD Group
Biological: Rabies vaccine — Participants will receive intramuscular injection of rabies vaccine (0.1 ml).
  Arms: Control Group

SUMMARY:
The study intends to establish proof of concept for a fractional dose schedule under conditions of natural exposure in children 5-17 months old at first vaccination. The study also aims to establish the role of third dose spacing in a fractional dose schedule, describe the effect of an earlier full fourth dose at Month 14 and describe the effect of multiple fractional or full yearly doses.

DETAILED DESCRIPTION:
The current study intends to establish proof of concept (POC) for a fractional dose schedule under conditions of natural exposure. The study will be conducted in children 5-17 months old at first vaccination living in areas of mid to high malaria transmission, in line with the age group recommended by the World Health Organization (WHO) for the implementation of the RTS,S/AS01E vaccine. Results from this study will be critical in informing future possibilities for the development of vaccine-based strategies which, in combination with other interventions, may contribute to the malaria elimination agenda.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. return for follow-up visits).
* Signed or thumb-printed and witnessed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by an independent witness.
* A male or female between, and including, five and 17 months of age at the time of the first vaccination.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* Previously received three documented doses of diphtheria, tetanus, pertussis, hepatitis B vaccine (DTPHepB), and at least three doses of oral polio vaccine.

Exclusion Criteria:

* Child in care.
* Use of a drug or vaccine that is not approved for that indication (by one of the following regulatory authorities: Food and Drug Administration [FDA; USA] or European Union member state or WHO [with respect to prequalification]) other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone (0.5 mg/kg/day (for pediatric participants) or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting seven days before each dose and ending seven days after each dose of vaccine administration.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of anaphylaxis post-vaccination.
* History of any, or documented, serious adverse reaction to rabies vaccination.
* Contraindication to rabies vaccination (Rabipur is contraindicated in participants with history of a severe hypersensitivity to any of the ingredients in the vaccine. Note that the vaccine contains polygeline and residues of chicken proteins, and may contain traces of neomycin, chlortetracycline and amphotericin B).
* Major congenital defects.
* Serious chronic illness.
* Children with a past history of a neurological disorder or atypical febrile seizure (a febrile seizure is atypical if it meets one of the following criteria: not associated with fever; lasts > 5 minutes; focal (not generalized); followed by transient or persistent neurological abnormality; occurs in a child < 6 months of age).
* Acute disease and/or fever at the time of enrolment. Fever is defined as temperature ≥ 37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route.

Participants with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.

* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Moderate or severe malnutrition at screening defined as weight for age or weight for height Z-score < -2.
* Hemoglobin concentration < 8 g/dl at screening.
* Same sex twins (to avoid misidentification).
* Maternal death.
* Prior receipt of an investigational malaria vaccine.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Kumasi, Ghana
- GSK Investigational Site, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Westercamp N, Osei-Tutu L, Schuerman L, Kariuki SK, Bollaerts A, Lee CK, Samuels AM, Ockenhouse C, Bii DK, Adjei S, Oneko M, Lievens M, Attobrah Sarfo MA, Atieno C, Bakari A, Sang T, Kotoh-Mortty MF, Otieno K, Roman F, Buabeng PBY, Ntiamoah Y, Ansong D, Agbenyega T, Ofori-Anyinam O. Could Less Be More? Accounting for Fractional-Dose Regimens and Different Number of Vaccine Doses When Measuring the Impact of the RTS,S/AS01E Malaria Vaccine. J Infect Dis. 2024 Aug 16;230(2):e486-e495. doi: 10.1093/infdis/jiae075. PMID 38438123
- [Derived] Osei-Tutu L, Kariuki SK, Lee CK, Fabre R, Bii DK, Adjei S, Oneko M, Attobrah Sarfo MA, Ockenhouse CF, Schuerman L, Buabeng PBY, Bakari A, Atieno C, Kotoh-Mortty MF, Otieno K, Ntiamoah Y, Sang T, Bollaerts A, Westercamp N, Ansong D, Agbenyega T, Samuels AM, Ofori-Anyinam O; RTS,S study group. Sustained efficacy of the RTS,S/AS01E malaria vaccine over 50 months of follow-up when used in full-dose or fractional-dose regimens in young children in Ghana and Kenya: final results from an open-label, phase 2b, randomised controlled trial. Lancet Glob Health. 2025 Oct;13(10):e1723-e1736. doi: 10.1016/S2214-109X(25)00272-4. PMID 40975080
- [Derived] Juraska M, Early AM, Li L, Schaffner SF, Lievens M, Khorgade A, Simpkins B, Hejazi NS, Benkeser DA, Wang Q, Mercer LD, Adjei S, Agbenyega T, Anderson S, Ansong D, Bii DK, Buabeng PBY, English S, Fitzgerald N, Grimsby J, Kariuki SK, Otieno K, Roman F, Samuels AM, Westercamp N, Ockenhouse CF, Ofori-Anyinam O, Lee CK, MacInnis BL, Wirth DF, Gilbert PB, Neafsey DE. Baseline malaria infection status and RTS,S/AS01E malaria vaccine efficacy. medRxiv [Preprint]. 2023 Nov 23:2023.11.22.23298907. doi: 10.1101/2023.11.22.23298907. PMID 38045387
- [Derived] Samuels AM, Ansong D, Kariuki SK, Adjei S, Bollaerts A, Ockenhouse C, Westercamp N, Lee CK, Schuerman L, Bii DK, Osei-Tutu L, Oneko M, Lievens M, Attobrah Sarfo MA, Atieno C, Morelle D, Bakari A, Sang T, Jongert E, Kotoh-Mortty MF, Otieno K, Roman F, Buabeng PBY, Ntiamoah Y, Ofori-Anyinam O, Agbenyega T; RTS,S study group. Efficacy of RTS,S/AS01E malaria vaccine administered according to different full, fractional, and delayed third or early fourth dose regimens in children aged 5-17 months in Ghana and Kenya: an open-label, phase 2b, randomised controlled trial. Lancet Infect Dis. 2022 Sep;22(9):1329-1342. doi: 10.1016/S1473-3099(22)00273-0. Epub 2022 Jun 23. PMID 35753316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As pre-specified in statistical analysis plan, data reported in Participant Flow, Baseline Characteristics and Adverse Events were presented for individual groups (R012-20 Group, R012-14-mD Group, R012-14-mD Group, Fx017-mFxD Group and Control Group).
Pre-assignment Details: As pre-specified in protocol, efficacy outcome measures corresponding to clinical malaria (primary case definition) and Plasmodium (P.) falciparum infection, presented data for R012-20+R012-14 Group (Pooled group) because the interventional strategy (1st dose at Month 0, 2nd dose at Month 1, 3rd dose at Month 2) was the same for both the R012-20 group and the R012-14 group until Month 14.
Groups:
- R012-20 Group: Participants received a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2 and at Month 20.
- R012-14-mD Group: Participants received a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2 and yearly full doses at Month 14, Month 26 and Month 38.
- Fx012-14-mFxD Group: Participants received a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 2 and yearly fractional doses at Month 14, Month 26 and Month 38.
- Fx017-mFxD Group: Participants received a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 7 and yearly fractional doses at Month 20 and Month 32.
- Control Group: Participants received rabies vaccine at Month 0, Month 1 and Month 2.
Period: Overall Study
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Started | 298 | 294 | 304 | 311 | 293
Completed | 229 | 232 | 242 | 247 | 237
Not Completed | 69 | 62 | 62 | 64 | 56
Not completed — Serious Adverse Event And/Or Pimd | 2 | 1 | 0 | 4 | 1
Not completed — Protocol Deviation | 2 | 0 | 1 | 2 | 1
Not completed — Consent Withdrawal, Not Due To An Adverse Event/A Serious Adverse Event | 29 | 21 | 13 | 21 | 16
Not completed — Migrated / Moved From The Study Area | 26 | 28 | 44 | 29 | 27
Not completed — Lost to Follow-up | 10 | 10 | 4 | 6 | 10
Not completed — Other | 0 | 2 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group | Total
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293 | 1500
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.2 (3.9) | 10.3 (3.8) | 10.5 (4.0) | 10.2 (3.8) | 10.5 (3.9) | 10.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 155 | 172 | 163 | 152 | 761
  Male | 179 | 139 | 132 | 148 | 141 | 739
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 298 | 294 | 304 | 311 | 293 | 1500

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Malaria Meeting the Primary Case Definition
Description: The primary case definition is: Plasmodium (P.) falciparum asexual parasitemia greater than (>)5000 parasites/microliters (μl) and presence of fever (axillary temperature greater than or equal to [≥]37.5°C) at the time of presentation and occurring in a child who is unwell and brought for treatment to a healthcare facility. The incidence is expressed as a person year rate for each group (n/T), representing the number of events (n) reported over the risk period, which was counted in days and expressed as person years at risk (T). The objective of this endpoint was to demonstrate the superiority of a Fx012-14-mFxD Group compared to a standard schedule of RTS,S/AS01E with three full doses (R012-20+R012-14 Group) in terms of vaccine efficacy. This analysis was reported for the R012-20+R012-14 Group (Pooled group) because the interventional strategy (1st dose at Month 0, 2nd dose at Month 1, 3rd dose at Month 2) was the same for both the R012-20 group and the R012-14 group until Month 14.
Time Frame: From Month 2.5 to Month 14
Population: This analysis was performed on Per Protocol Set (PPS) for efficacy, which included all participants from Exposed Set (ES) who fulfilled eligibility criteria and received all interventions as per study plan, within the protocol specified intervals that contribute to the time at risk in the follow-up period starting Month 2.5 to Month 14. As pre-specified in the analysis plan, the analysis of this outcome measure was reported for the R012-20+R012-14 Group and the Fx012-14-mFxD Group.
Measure: Number; unit: events per person-year
Groups:
- R012-20 + R012-14 Group: Participants received full doses of RTS,S/AS01E at Month 0, Month 1, Month 2 and a full dose at Month 14, Month 20, Month 26, Month 38.
Arm/Group | Fx012-14-mFxD Group | R012-20 + R012-14 Group
Number analyzed (Participants) | 271 | 523
events per person-year | 0.45 | 0.36
Statistical Analysis 1: Comparison: Fx012-14-mFxD Group vs R012-20 + R012-14 Group; To demonstrate the superiority of a 3-dose schedule of GSK Biologicals' malaria vaccine RTS,S/AS01E with a fractional third dose at Month 2 (Fx012-14-mFxD Group) compared to a standard schedule of RTS,S/AS01E with 3 full doses (R012-20 + R012-14 Group) in terms of vaccine efficacy against clinical malaria (primary case definition) over 12 months post-Dose 3; Test type: Superiority; p = 0.154, Regression, Cox; The 95% Confidence Interval of the incremental vaccine efficacy estimates was calculated from Cox regression model; Incremental vaccine efficacy = -21, 95% CI 2-sided [-57 to 7]

2. Secondary Outcome: Incidence of Clinical Malaria Meeting the Primary and Secondary Case Definitions of the Fx012-14-mFxD Group Versus the R012-20 Group
Description: The primary case definition is P. falciparum asexual parasitemia > 5000 μl and presence of fever (axillary temperature ≥ 37.5°C) at the time of presentation and occurring in a child who is unwell and brought for treatment to a healthcare facility.
  The secondary case definition is P. falciparum asexual parasitemia > 0 and presence of fever (axillary temperature ≥ 37.5°C) at the time of presentation or history of fever within 24 hours of presentation and occurring in a child who is unwell and brought for treatment to a healthcare facility. The incidence of clinical malaria for primary and secondary case definition is expressed as n/T, representing the n reported over the risk period, which was counted in days and expressed as T.
Time Frame: From Month 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine. As per statistical analysis plan, the analysis of this outcome measure was reported only for the Fx012-14-mFxD Group and the R012-20 Group since the objective of this endpoint was to assess the vaccine efficacy in terms of incident rate against Fx012-14-mFxD Group versus R012-20 Group.
Measure: Number; unit: events per person-year
Arm/Group | Fx012-14-mFxD Group | R012-20 Group
Number analyzed (Participants) | 304 | 298
events per person-year
  Primary case definition | 0.69 | 0.86
  Secondary case definition | 1.18 | 1.62

3. Secondary Outcome: Incidence of Clinical Malaria Meeting the Primary and Secondary Case Definitions of the Fx012-14-mFxD Group Versus the R012-14-mD Group
Description: as for outcome 2
Time Frame: From Month 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine. As per statistical analysis plan, the analysis of this outcome measure was reported only for the Fx012-14-mFxD Group and the R012-14-mD Group since the objective of this endpoint was to assess the vaccine efficacy in terms of incident rate against Fx012-14-mFxD Group versus R012-14-mD Group..
Measure: Number; unit: events per person-year
Arm/Group | Fx012-14-mFxD Group | R012-14-mD Group
Number analyzed (Participants) | 304 | 294
events per person-year
  Primary case definition | 0.69 | 0.67
  Secondary case definition | 1.18 | 1.22

4. Secondary Outcome: The Prevalence of P. Falciparum Infections Defined by Positive Blood Slide at Each Cross-sectional Survey
Description: Prevalence of P. falciparum infections of each RTS,S/AS01E schedule at cross-sectional visits. As specified in the statistical analysis plan, a graphical presentation of the prevalence over time was analyzed for this outcome measure and only the percentage values were reported to depict the prevalence of P. falciparum infections.
Time Frame: Monthly from Month 0 to Month 20 and every 3 months thereafter until Study End (Month 50)
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine and for whom data were assessed during specific timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Percentage of participants
  Month 0 | 10.1 | 6.1 | 4.6 | 5.1 | 7.2
  Month 1 | 3.8 | 5.9 | 3.1 | 5.7 | 5.7
  Month 2 | 4.3 | 4.6 | 2.8 | 5.5 | 3.9
  Month 3 | 3.0 | 4.1 | 3.2 | 6.5 | 5.4
  Month 4 | 3.9 | 4.7 | 2.3 | 4.9 | 5.6
  Month 5 | 3.9 | 3.6 | 1.9 | 4.7 | 8.5
  Month 6 | 4.8 | 4.4 | 3.0 | 6.2 | 7.2
  Month 7 | 6.0 | 7.7 | 6.5 | 5.3 | 4.8
  Month 8 | 4.0 | 7.2 | 5.0 | 4.4 | 9.4
  Month 9 | 6.7 | 6.6 | 6.8 | 7.1 | 9.7
  Month 10 | 6.0 | 5.3 | 7.4 | 6.7 | 12.7
  Month 11 | 8.4 | 5.7 | 6.9 | 7.8 | 12.5
  Month 12 | 9.7 | 6.5 | 6.9 | 6.6 | 13.1
  Month 13 | 7.3 | 6.9 | 7.7 | 9.7 | 13.5
  Month 14 | 12.6 | 2.0 | 5.3 | 7.1 | 12.9
  Month 15 | 8.3 | 3.7 | 5.1 | 6.4 | 9.0
  Month 16 | 7.9 | 6.7 | 6.8 | 5.7 | 6.7
  Month 17 | 10.8 | 9.8 | 7.0 | 5.7 | 11.7
  Month 18 | 9.3 | 9.9 | 7.1 | 6.5 | 12.2
  Month 19 | 6.8 | 7.9 | 8.8 | 9.7 | 10.1
  Month 20 | 7.0 | 8.3 | 8.1 | 3.4 | 7.5
  Month 23 | 11.3 | 7.3 | 11.2 | 7.5 | 10.7
  Month 26 | 12.2 | 2.8 | 6.0 | 9.5 | 10.9
  Month 29 | 10.6 | 6.9 | 9.2 | 8.7 | 13.4
  Month 32 | 10.5 | 7.9 | 7.9 | 5.8 | 10.6
  Month 35 | 10.9 | 11.0 | 10.1 | 10.4 | 13.7
  Month 38 | 11.5 | 6.5 | 7.3 | 8.4 | 17.0
  Month 41 | 5.8 | 7.5 | 6.8 | 6.5 | 11.0
  Month 44 | 12.3 | 10.2 | 9.8 | 8.7 | 11.9
  Month 47 | 13.8 | 5.7 | 8.9 | 8.3 | 16.2
  Month 50 | 13.1 | 10.8 | 13.6 | 12.6 | 13.5

5. Secondary Outcome: Incidence of P. Falciparum Infections Defined by Positive Blood Slide
Description: The incidence of P. falciparum infections is expressed as n/T, representing the n reported over the risk period, which was counted in days and expressed as T.
  Assessment of vaccine efficacy (VE) against first or only episodes of incident P. falciparum infections defined by positive blood slide over the entire study period (Month 0 to Month 50) was not done after the Month 21 Interim analysis since it was assumed that almost all children would have already contracted malaria at least once.
Time Frame: Month 0 to Month 14
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine and for whom data were collected from Month 0 to Month 14. As pre-specified in the analysis plan, the analysis of the outcome measure was reported for the R012-20+R012-14 Group (Pooled group) because the interventional strategy (1st dose at Month 0, 2nd dose at Month 1 and 3rd dose at Month 2) was the same for both the R012-20 group and the R012-14 group until Month 14.
Measure: Number; unit: events per person-year
Arm/Group | R012-20 + R012-14 Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 543 | 290 | 295 | 272
events per person-year | 0.50 | 0.60 | 0.59 | 0.80

6. Secondary Outcome: Number of Seropositive Participants for Anti-circumsporozoite (Anti-CS) Antibodies
Description: A seropositive participant is defined as a participant with antibody concentrations ≥ 0.5 ELISA units per milliliter (EU/mL).
Time Frame: Before Dose 1, one month post-Dose 2, before and one month post-Dose 3, before and one month after Dose 4, before and one month after each yearly dose and at Study End (Month 50)
Population: The analysis was performed on immunosubset which included all participants who complied with protocol defined procedures and for whom immunogenicity results were available for the specified time point and specific assay.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 45 | 49 | 45 | 49 | 48
Participants
  Before Dose 1, Pre-Vaccination (Day 1) | 2 | 1 | 0 | 2 | 2
  Post Dose 2 (Month 2): number analyzed (Participants) | 43 | 48 | 42 | 48 | 46
  Post Dose 2 (Month 2) | 43 | 48 | 42 | 47 | 4
  Post Dose 3 (Month 3): number analyzed (Participants) | 36 | 44 | 41 | 0 | 43
  Post Dose 3 (Month 3) | 36 | 44 | 40 |  | 2
  Pre-Dose 3 (Month 7): number analyzed (Participants) | 0 | 0 | 0 | 44 | 0
  Pre-Dose 3 (Month 7) |  |  |  | 44 |
  Post Dose 3 (Month 8): number analyzed (Participants) | 0 | 0 | 0 | 43 | 0
  Post Dose 3 (Month 8) |  |  |  | 43 |
  Pre-Dose 4 (Month 14): number analyzed (Participants) | 0 | 42 | 40 | 0 | 0
  Pre-Dose 4 (Month 14) |  | 41 | 40 |  |
  Post Dose 4 (Month 15): number analyzed (Participants) | 0 | 37 | 38 | 0 | 0
  Post Dose 4 (Month 15) |  | 37 | 38 |  |
  Pre-Dose 4 (Month 20): number analyzed (Participants) | 37 | 0 | 0 | 42 | 37
  Pre-Dose 4 (Month 20) | 37 |  |  | 42 | 2
  Post Dose 4 (Month 21): number analyzed (Participants) | 35 | 0 | 0 | 39 | 0
  Post Dose 4 (Month 21) | 35 |  |  | 39 |
  Pre-Dose 5 (Month 26): number analyzed (Participants) | 0 | 38 | 34 | 0 | 0
  Pre-Dose 5 (Month 26) |  | 37 | 34 |  |
  Post Dose 5 (Month 27): number analyzed (Participants) | 0 | 30 | 26 | 0 | 0
  Post Dose 5 (Month 27) |  | 30 | 26 |  |
  Pre-Dose 5 (Month 32): number analyzed (Participants) | 0 | 0 | 0 | 37 | 0
  Pre-Dose 5 (Month 32) |  |  |  | 37 |
  Post Dose 5 (Month 33): number analyzed (Participants) | 0 | 0 | 0 | 32 | 0
  Post Dose 5 (Month 33) |  |  |  | 32 |
  Pre-Dose 6 (Month 38): number analyzed (Participants) | 0 | 34 | 31 | 0 | 0
  Pre-Dose 6 (Month 38) |  | 34 | 31 |  |
  Post Dose 6 (Month 39): number analyzed (Participants) | 0 | 33 | 28 | 0 | 0
  Post Dose 6 (Month 39) |  | 33 | 28 |  |
  End of Study (Month 50): number analyzed (Participants) | 30 | 34 | 29 | 25 | 37
  End of Study (Month 50) | 30 | 34 | 29 | 25 | 2

7. Secondary Outcome: Number of Seropositive Participants for Anti-hepatitis B (Anti-HB) Antibodies
Description: A seropositive participant is defined as a participant with antibody concentrations ≥ 10 milli-international units per milliliter (mIU/mL).
Time Frame: as for outcome 6
Population: The analysis was performed on the immunosubset which included all participants who complied with protocol defined procedures and for whom immunogenicity results were available for the specified time point and specific assay.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 45 | 49 | 44 | 48 | 48
Participants
  Before Dose 1, Pre-Vaccination (Day 1) | 42 | 48 | 39 | 40 | 43
  Post Dose 2 (Month 2): number analyzed (Participants) | 43 | 48 | 41 | 48 | 48
  Post Dose 2 (Month 2) | 43 | 48 | 41 | 48 | 42
  Post Dose 3 (Month 3): number analyzed (Participants) | 35 | 44 | 40 | 0 | 43
  Post Dose 3 (Month 3) | 35 | 44 | 40 |  | 39
  Pre-Dose 3 (Month 7): number analyzed (Participants) | 0 | 0 | 0 | 44 | 0
  Pre-Dose 3 (Month 7) |  |  |  | 44 |
  Post Dose 3 (Month 8): number analyzed (Participants) | 0 | 0 | 0 | 43 | 0
  Post Dose 3 (Month 8) |  |  |  | 43 |
  Pre-Dose 4 (Month 14): number analyzed (Participants) | 0 | 41 | 40 | 0 | 0
  Pre-Dose 4 (Month 14) |  | 41 | 40 |  |
  Post Dose 4 (Month 15): number analyzed (Participants) | 0 | 37 | 37 | 0 | 0
  Post Dose 4 (Month 15) |  | 37 | 37 |  |
  Pre-Dose 4 (Month 20): number analyzed (Participants) | 37 | 0 | 0 | 42 | 37
  Pre-Dose 4 (Month 20) | 37 |  |  | 42 | 30
  Post Dose 4 (Month 21): number analyzed (Participants) | 33 | 0 | 0 | 38 | 0
  Post Dose 4 (Month 21) | 33 |  |  | 38 |
  Pre-Dose 5 (Month 26): number analyzed (Participants) | 0 | 38 | 34 | 0 | 0
  Pre-Dose 5 (Month 26) |  | 38 | 34 |  |
  Post Dose 5 (Month 27): number analyzed (Participants) | 0 | 30 | 26 | 0 | 0
  Post Dose 5 (Month 27) |  | 30 | 26 |  |
  Pre-Dose 5 (Month 32): number analyzed (Participants) | 0 | 0 | 0 | 37 | 0
  Pre-Dose 5 (Month 32) |  |  |  | 37 |
  Post Dose 5 (Month 33): number analyzed (Participants) | 0 | 0 | 0 | 32 | 0
  Post Dose 5 (Month 33) |  |  |  | 32 |
  Pre-Dose 6 (Month 38): number analyzed (Participants) | 0 | 34 | 31 | 0 | 0
  Pre-Dose 6 (Month 38) |  | 34 | 31 |  |
  Post Dose 6 (Month 39): number analyzed (Participants) | 0 | 33 | 28 | 0 | 0
  Post Dose 6 (Month 39) |  | 33 | 28 |  |
  End of Study (Month 50): number analyzed (Participants) | 30 | 34 | 28 | 25 | 36
  End of Study (Month 50) | 30 | 34 | 28 | 25 | 22

8. Secondary Outcome: Antibody Concentrations for Anti-CS
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as EU/mL.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 45 | 49 | 45 | 49 | 48
EU/mL
  Before Dose 1, Pre-Vaccination (Day 1) | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.0]
  Post Dose 2 (Month 2): number analyzed (Participants) | 43 | 48 | 42 | 48 | 46
  Post Dose 2 (Month 2) | 359.9 [284.3 to 455.5] | 320.0 [248.2 to 412.6] | 378.8 [279.3 to 513.9] | 253.6 [182.2 to 353.0] | 1.3 [0.9 to 1.9]
  Post Dose 3 (Month 3): number analyzed (Participants) | 36 | 44 | 41 | 0 | 43
  Post Dose 3 (Month 3) | 472.6 [371.0 to 602.0] | 342.5 [275.6 to 425.6] | 251.1 [170.6 to 369.6] |  | 1.0 [0.9 to 1.1]
  Pre-Dose 3 (Month 7): number analyzed (Participants) | 0 | 0 | 0 | 44 | 0
  Pre-Dose 3 (Month 7) |  |  |  | 25.3 [19.1 to 33.5] |
  Post Dose 3 (Month 8): number analyzed (Participants) | 0 | 0 | 0 | 43 | 0
  Post Dose 3 (Month 8) |  |  |  | 142.3 [113.9 to 177.8] |
  Pre-Dose 4 (Month 14): number analyzed (Participants) | 0 | 42 | 40 | 0 | 0
  Pre-Dose 4 (Month 14) |  | 26.9 [19.2 to 37.7] | 22.6 [17.9 to 28.5] |  |
  Post Dose 4 (Month 15): number analyzed (Participants) | 0 | 37 | 38 | 0 | 0
  Post Dose 4 (Month 15) |  | 234.8 [184.2 to 299.5] | 196.4 [150.4 to 256.7] |  |
  Pre-Dose 4 (Month 20): number analyzed (Participants) | 37 | 0 | 0 | 42 | 37
  Pre-Dose 4 (Month 20) | 26.6 [19.1 to 37.0] |  |  | 33.3 [23.5 to 47.3] | 1.0 [0.9 to 1.2]
  Post Dose 4 (Month 21): number analyzed (Participants) | 35 | 0 | 0 | 39 | 0
  Post Dose 4 (Month 21) | 288.1 [227.7 to 364.4] |  |  | 187.1 [139.9 to 250.1] |
  Pre-Dose 5 (Month 26): number analyzed (Participants) | 0 | 38 | 34 | 0 | 0
  Pre-Dose 5 (Month 26) |  | 37.3 [26.7 to 52.3] | 38.0 [27.7 to 52.1] |  |
  Post Dose 5 (Month 27): number analyzed (Participants) | 0 | 30 | 26 | 0 | 0
  Post Dose 5 (Month 27) |  | 185.2 [140.4 to 244.3] | 145.6 [106.6 to 198.9] |  |
  Pre-Dose 5 (Month 32): number analyzed (Participants) | 0 | 0 | 0 | 37 | 0
  Pre-Dose 5 (Month 32) |  |  |  | 38.9 [27.6 to 54.9] |
  Post Dose 5 (Month 33): number analyzed (Participants) | 0 | 0 | 0 | 32 | 0
  Post Dose 5 (Month 33) |  |  |  | 133.9 [103.4 to 173.4] |
  Pre-Dose 6 (Month 38): number analyzed (Participants) | 0 | 34 | 31 | 0 | 0
  Pre-Dose 6 (Month 38) |  | 45.7 [33.5 to 62.2] | 40.5 [31.0 to 52.9] |  |
  Post Dose 6 (Month 39): number analyzed (Participants) | 0 | 33 | 28 | 0 | 0
  Post Dose 6 (Month 39) |  | 181.8 [137.2 to 241.0] | 115.2 [86.4 to 153.6] |  |
  End of Study (Month 50): number analyzed (Participants) | 30 | 34 | 29 | 25 | 37
  End of Study (Month 50) | 25.1 [18.8 to 33.6] | 49.7 [37.0 to 66.6] | 35.5 [27.2 to 46.5] | 30.9 [19.9 to 47.9] | 1.0 [0.9 to 1.2]

9. Secondary Outcome: Antibody Concentrations for Anti-HB
Description: The antibody concentrations were calculated as GMCs and expressed as mlU/mL.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mlU/mL
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 45 | 49 | 44 | 48 | 48
mlU/mL
  Before Dose 1, Pre-Vaccination (Day 1) | 162.8 [98.7 to 268.5] | 224.7 [142.3 to 354.7] | 124.6 [72.0 to 215.5] | 98.4 [55.7 to 173.8] | 152.5 [93.4 to 249.0]
  Post Dose 2 (Month 2): number analyzed (Participants) | 43 | 48 | 41 | 48 | 46
  Post Dose 2 (Month 2) | 39990.7 [23198.3 to 68938.5] | 39336.5 [26109.5 to 59264.5] | 34301.2 [19896.6 to 59134.2] | 29015.8 [17445.6 to 48259.4] | 159.1 [83.8 to 302.2]
  Post Dose 3 (Month 3): number analyzed (Participants) | 35 | 44 | 40 | 0 | 43
  Post Dose 3 (Month 3) | 45665.7 [26775.1 to 77884.4] | 37592.9 [27463.3 to 51458.8] | 21641.4 [12408.6 to 37743.9] |  | 100.4 [57.3 to 175.7]
  Pre-Dose 3 (Month 7): number analyzed (Participants) | 0 | 0 | 0 | 44 | 0
  Pre-Dose 3 (Month 7) |  |  |  | 6296.7 [3817.3 to 10386.7] |
  Post Dose 3 (Month 8): number analyzed (Participants) | 0 | 0 | 0 | 43 | 0
  Post Dose 3 (Month 8) |  |  |  | 53700.6 [38222.8 to 75446.0] |
  Pre-Dose 4 (Month 14): number analyzed (Participants) | 0 | 41 | 40 | 0 | 0
  Pre-Dose 4 (Month 14) |  | 5700.6 [4033.4 to 8057.1] | 4856.5 [3129.3 to 7537.0] |  |
  Post Dose 4 (Month 15): number analyzed (Participants) | 0 | 37 | 37 | 0 | 0
  Post Dose 4 (Month 15) |  | 137582.9 [108671.7 to 174185.8] | 81612.1 [60532.7 to 110032.1] |  |
  Pre-Dose 4 (Month 20): number analyzed (Participants) | 37 | 0 | 0 | 42 | 37
  Pre-Dose 4 (Month 20) | 5189.6 [3061.3 to 8797.4] |  |  | 9700.1 [6732.0 to 13977.0] | 45.6 [26.6 to 78.3]
  Post Dose 4 (Month 21): number analyzed (Participants) | 33 | 0 | 0 | 38 | 0
  Post Dose 4 (Month 21) | 210277.6 [160964.7 to 274697.9] |  |  | 74185.9 [55296.5 to 99528.0] |
  Pre-Dose 5 (Month 26): number analyzed (Participants) | 0 | 38 | 34 | 0 | 0
  Pre-Dose 5 (Month 26) |  | 18767.8 [14581.3 to 24156.3] | 14130.8 [9985.9 to 19996.1] |  |
  Post Dose 5 (Month 27): number analyzed (Participants) | 0 | 30 | 26 | 0 | 0
  Post Dose 5 (Month 27) |  | 126992.7 [101650.7 to 158652.5] | 63683.7 [42424.1 to 95596.9] |  |
  Pre-Dose 5 (Month 32): number analyzed (Participants) | 0 | 0 | 0 | 37 | 0
  Pre-Dose 5 (Month 32) |  |  |  | 13212.6 [9396.3 to 18579.0] |
  Post Dose 5 (Month 33): number analyzed (Participants) | 0 | 0 | 0 | 32 | 0
  Post Dose 5 (Month 33) |  |  |  | 57655.7 [44884.3 to 74060.9] |
  Pre-Dose 6 (Month 38): number analyzed (Participants) | 0 | 34 | 31 | 0 | 0
  Pre-Dose 6 (Month 38) |  | 24027.2 [18417.3 to 31345.9] | 16776.6 [11990.4 to 23473.1] |  |
  Post Dose 6 (Month 39): number analyzed (Participants) | 0 | 33 | 28 | 0 | 0
  Post Dose 6 (Month 39) |  | 114277.1 [88950.0 to 146815.7] | 60669.1 [42343.5 to 86925.7] |  |
  End of Study (Month 50): number analyzed (Participants) | 30 | 34 | 28 | 25 | 36
  End of Study (Month 50) | 10714.9 [7199.2 to 15947.3] | 24353.9 [18411.6 to 32214.0] | 13240.2 [9550.0 to 18356.2] | 10013.0 [6511.4 to 15397.7] | 18.5 [10.4 to 32.8]

10. Secondary Outcome: Number of Participants With Any, Fatal and Related Serious Adverse Events (SAEs)
Description: SAEs assessed included any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related SAEs= Any SAE related to investigational vaccine or related to study participation or to a GSK concomitant medication/vaccine as assessed by the investigator. Fatal SAEs= Any SAEs leading to death.
Time Frame: From Day 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants
  Any SAE | 73 | 65 | 64 | 84 | 92
  Fatal SAE | 2 | 1 | 0 | 4 | 1
  Related SAE | 3 | 0 | 0 | 2 | 0

11. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and SAEs Leading to Withdrawal From Further Vaccination
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product.
  SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants | 2 | 1 | 0 | 4 | 1

12. Secondary Outcome: Number of Participants With Cerebral Malaria and Severe Malaria
Description: Cerebral malaria is defined as Severe P. falciparum malaria with coma (Blantyre coma score less than [<] 3); and if malaria with seizure: coma persisting for > 30 min after the seizure. Other treatable causes of coma should be excluded before diagnosing cerebral malaria (e.g. hypoglycaemia, bacterial meningitis).
  Severe malaria is defined as P. falciparum parasitemia > 0 detected by microscopy and/or rapid diagnostic test (RDT) and one or more of the following, occurring in the absence of an identified alternative cause: Impaired consciousness, Prostration, Multiple convulsions, Acidosis, Hypoglycemia, Severe malarial anemia, Renal impairment, Jaundice, Pulmonary edema, Significant bleeding: including recurrent or prolonged bleeding from the nose, gums or venipuncture sites, hematemesis or melaena, Shock, Hyperparasitemia.
Time Frame: From Day 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants
  Cerebral malaria | 0 | 0 | 0 | 0 | 1
  Severe malaria | 29 | 22 | 25 | 31 | 51

13. Secondary Outcome: Number of Participants With Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants | 0 | 2 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Meningitis
Description: Meningitis is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders.
Time Frame: From Day 0 to Month 50
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants | 1 | 1 | 1 | 3 | 3

15. Secondary Outcome: Number of Participants With Seizures
Description: Seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders.
Time Frame: During the 30-day (Day 0 to Day 29) follow-up period after any dose of study vaccine
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants | 5 | 1 | 0 | 4 | 4

16. Secondary Outcome: Number of Participants With Generalized Convulsive Seizures
Description: Generalized convulsive seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders.
Time Frame: During the 7-day (Day 0 to Day 6) follow-up period after any dose of study vaccine
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants | 4 | 1 | 0 | 4 | 2

17. Secondary Outcome: Number of Participants With Any Unsolicited AEs
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 30-day (Day 0 to Day 29) follow-up period following the 1st 3 doses and post dose 4, 5 and 6 of study vaccine
Population: The analysis was performed on ES which included all participants who received at least one dose of study vaccine and who had safety data available for the specific duration.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Participants
  Post 1st 3 doses | 223 | 221 | 240 | 242 | 238
  Post Dose 4: number analyzed (Participants) | 244 | 256 | 266 | 267 | 0
  Post Dose 4 | 74 | 94 | 101 | 79 |
  Post Dose 5: number analyzed (Participants) | 0 | 247 | 251 | 259 | 0
  Post Dose 5 |  | 67 | 65 | 88 |
  Post Dose 6: number analyzed (Participants) | 0 | 231 | 245 | 0 | 0
  Post Dose 6 |  | 64 | 76 |  |

18. Secondary Outcome: Number of Participants With Grade 4 Hematology and Biochemical Toxicities Before Dose 3
Description: The assessed parameters (alanine aminotransferase [ALT], creatinine, haemoglobin, white blood cells [WBC], platelets) were summarized according to DAIDS, 2004 (Division of AIDS). Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling. Data are presented for those participants who experienced Grade 4 toxicities. Grade 4 hematological toxicities included ALT: > 10.0 x ULN (Upper limit of normal), creatine: > 6.0 x ULN or requires dialysis, WBC: < 1.0 x 103 per microliter, platelets: < 25 x 103/μl and clinical signs of bleeding, and hemoglobin: < 5.0 grams/deciliter and clinical signs of heart failure.
Time Frame: Before Dose 3 (at Month 2)
Population: The analysis was performed on the reactogenicity sub-cohort, which included the first 50 participants enrolled in each group and for whom specific lab parameter data was available at a specific timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 46 | 48 | 44 | 45 | 49
Participants
  Haemoglobin | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0
  ALT | 0 | 0 | 0 | 0 | 0
  Creatine | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Grade 4 Hematology and Biochemical Toxicities at 7 Days Post-Dose 3
Description: The assessed parameters (ALT, creatinine, haemoglobin, WBC, platelets) were summarized according to DAIDS, 2004 (Division of AIDS). Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling. Data are presented for those participants who experienced Grade 4 toxicities. Grade 4 hematological toxicities included ALT: > 10.0 x ULN, creatine: > 6.0 x ULN or requires dialysis, WBC: < 1.0 x 103 per microliter, platelets: < 25 x 103/μl and clinical signs of bleeding, and hemoglobin: < 5.0 grams/deciliter and clinical signs of heart failure.
Time Frame: At 7 days post-Dose 3
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 44 | 47 | 43 | 41 | 48
Participants
  Haemoglobin | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0
  ALT | 0 | 0 | 0 | 0 | 0
  Creatine | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Grade 4 Hematology and Biochemical Toxicities at 30 Days Post-Dose 3
Description: as for outcome 19
Time Frame: At 30 days post-Dose 3
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 38 | 45 | 42 | 44 | 49
Participants
  Haemoglobin | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0
  ALT | 0 | 0 | 0 | 0 | 0
  Creatine | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Any Solicited Local Symptoms
Description: Assessed solicited local AEs are: redness, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade. Any redness and swelling = adverse event reported with a surface diameter > 0 millimeters.
Time Frame: During the 4-day (Day 0 to Day 3) follow-up period after Dose 3, Dose 4, Dose 5 and Dose 6 of study vaccination
Population: The analysis was performed on Solicited Safety Set reactogenicity sub-cohort (SSRS) which included all participants who received at least one dose of study vaccine and had solicited local data during specific duration.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 46 | 48 | 44 | 45 | 49
Participants
  Any Erythema, after Dose 3 | 0 | 1 | 0 | 0 | 0
  Any Erythema, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Erythema, after Dose 4 | 0 | 0 | 0 | 0 |
  Any Erythema, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Erythema, after Dose 5 |  | 0 | 0 | 0 |
  Any Erythema, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Erythema, after Dose 6 |  | 0 | 0 |  |
  Any Pain, after Dose 3 | 1 | 1 | 0 | 0 | 0
  Any Pain, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Pain, after Dose 4 | 1 | 1 | 0 | 4 |
  Any Pain, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Pain, after Dose 5 |  | 4 | 1 | 0 |
  Any Pain, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Pain, after Dose 6 |  | 3 | 0 |  |
  Any Swelling, after Dose 3 | 0 | 1 | 0 | 1 | 0
  Any Swelling, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Swelling, after Dose 4 | 1 | 0 | 0 | 1 |
  Any Swelling, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Swelling, after Dose 5 |  | 0 | 1 | 1 |
  Any Swelling, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Swelling, after Dose 6 |  | 0 | 0 |  |

22. Secondary Outcome: Number of Participants With Any Solicited General Symptoms
Description: Assessed solicited general AEs are: drowsiness, irritability/fussiness and loss of appetite. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
Time Frame: During the 4-day (Day 0 to Day 3) follow-up period after Dose 3, Dose 4, Dose 5 and Dose 6 of study vaccination
Population: The analysis was performed on SSRS which included all participants who received at least one dose of study vaccine and had solicited general data during specific duration.
Measure: Count of Participants; unit: Participants
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 46 | 48 | 44 | 45 | 49
Participants
  Any Drowsiness, after Dose 3 | 2 | 0 | 1 | 2 | 0
  Any Drowsiness, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Drowsiness, after Dose 4 | 0 | 2 | 1 | 0 |
  Any Drowsiness, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Drowsiness, after Dose 5 |  | 0 | 1 | 0 |
  Any Drowsiness, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Drowsiness, after Dose 6 |  | 0 | 0 |  |
  Any Irritability/Fussiness, after Dose 3 | 0 | 1 | 0 | 3 | 0
  Any Irritability/Fussiness, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Irritability/Fussiness, after Dose 4 | 0 | 6 | 0 | 1 |
  Any Irritability/Fussiness, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Irritability/Fussiness, after Dose 5 |  | 0 | 0 | 0 |
  Any Irritability/Fussiness, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Irritability/Fussiness, after Dose 6 |  | 0 | 0 |  |
  Any Loss of appetite, after Dose 3 | 0 | 1 | 0 | 1 | 0
  Any Loss of appetite, after Dose 4: number analyzed (Participants) | 41 | 44 | 42 | 43 | 0
  Any Loss of appetite, after Dose 4 | 2 | 5 | 2 | 0 |
  Any Loss of appetite, after Dose 5: number analyzed (Participants) | 0 | 42 | 39 | 43 | 0
  Any Loss of appetite, after Dose 5 |  | 0 | 1 | 0 |
  Any Loss of appetite, after Dose 6: number analyzed (Participants) | 0 | 39 | 38 | 0 | 0
  Any Loss of appetite, after Dose 6 |  | 0 | 0 |  |

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Month 0 to Month 50. All-Cause Mortality: From Month 0 to Month 50. Other Adverse Events: Solicited Adverse Events were collected during the 4-day follow-up period after vaccination and Unsolicited Adverse Events during the 30-day follow-up period after vaccination
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/298 | 1/294 | 0/304 | 4/311 | 1/293
Serious Adverse Events (participants affected / at risk) | 73/298 | 65/294 | 64/304 | 84/311 | 92/293
Other Adverse Events (participants affected / at risk) | 230/298 | 243/294 | 253/304 | 253/311 | 234/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R012-20 Group (N=298) | R012-14-mD Group (N=294) | Fx012-14-mFxD Group (N=304) | Fx017-mFxD Group (N=311) | Control Group (N=293)
Plasmodium falciparum infection (Infections and infestations) | 28 (28) | 22 (22) | 29 (29) | 32 (32) | 48 (48)
Pneumonia (Infections and infestations) | 15 (15) | 15 (15) | 12 (12) | 10 (10) | 21 (21)
Gastroenteritis (Infections and infestations) | 12 (12) | 9 (9) | 9 (9) | 15 (15) | 13 (13)
Malaria (Infections and infestations) | 8 (8) | 7 (7) | 6 (6) | 10 (10) | 12 (12)
Otitis media (Infections and infestations) | 4 (4) | 3 (3) | 4 (4) | 4 (4) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Meningitis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Otitis media acute (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Dysentery (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bullous impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoid abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis enteroviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 10 (10) | 4 (4) | 6 (6) | 12 (12) | 11 (11)
Seizure (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 4 (4) | 4 (4) | 11 (11)
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 5 (5)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in mouth (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R012-20 Group (N=298) | R012-14-mD Group (N=294) | Fx012-14-mFxD Group (N=304) | Fx017-mFxD Group (N=311) | Control Group (N=293)
Upper respiratory tract infection (Infections and infestations) | 161 (238) | 187 (320) | 198 (377) | 194 (323) | 164 (237)
Malaria (Infections and infestations) | 76 (101) | 86 (142) | 98 (147) | 94 (142) | 63 (90)
Gastroenteritis (Infections and infestations) | 56 (65) | 87 (107) | 76 (95) | 70 (86) | 68 (80)
Pneumonia (Infections and infestations) | 19 (20) | 41 (44) | 38 (42) | 26 (28) | 33 (34)
Conjunctivitis (Infections and infestations) | 24 (26) | 32 (35) | 35 (37) | 22 (23) | 27 (28)
Otitis media (Infections and infestations) | 23 (25) | 25 (29) | 33 (37) | 21 (24) | 33 (38)
Skin bacterial infection (Infections and infestations) | 18 (20) | 25 (29) | 29 (35) | 16 (18) | 16 (18)
Respiratory tract infection (Infections and infestations) | 18 (19) | 15 (16) | 16 (16) | 10 (10) | 11 (11)
Rash pustular (Infections and infestations) | 9 (9) | 12 (12) | 11 (13) | 17 (18) | 11 (11)
Body tinea (Infections and infestations) | 4 (4) | 11 (12) | 11 (11) | 9 (9) | 11 (12)
Septic rash (Infections and infestations) | 10 (12) | 9 (11) | 10 (10) | 11 (11) | 2 (2)
Tinea capitis (Infections and infestations) | 8 (8) | 9 (10) | 8 (8) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 8 (9) | 7 (7) | 1 (1) | 6 (6)
Oral candidiasis (Infections and infestations) | 6 (6) | 5 (5) | 2 (3) | 1 (1) | 7 (7)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 4 (4) | 2 (2) | 3 (3)
Abscess (Infections and infestations) | 6 (6) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
Dysentery (Infections and infestations) | 2 (2) | 4 (4) | 5 (5) | 3 (3) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 3 (3) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 5 (5) | 3 (3) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Wound sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Helminthic infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 2 (2)
Furuncle (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cutaneous larva migrans (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bullous impetigo (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecthyma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taeniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 26 (27) | 30 (35) | 27 (28) | 22 (25) | 24 (25)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7) | 3 (3) | 8 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (10) | 3 (3) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 2 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Rash vesicular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 35 (41) | 69 (103) | 36 (43) | 43 (49) | 13 (14)
Injection site pain (General disorders) | 4 (4) | 9 (12) | 2 (2) | 4 (4) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 4 (5) | 1 (1) | 2 (3) | 0 (0)
Irritability postvaccinal (General disorders) | 0 (0) | 6 (7) | 0 (0) | 4 (4) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 30 (34) | 25 (26) | 40 (44) | 26 (30) | 35 (41)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3) | 7 (8) | 3 (3) | 5 (5)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 9 (9) | 10 (11) | 17 (19) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (8) | 12 (14) | 7 (8) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4) | 5 (5) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 7 (7) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Vernal keratoconjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03276962/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03276962/SAP_001.pdf